CLINICAL TRIAL: NCT06170684
Title: Clinical Study of Conservative Treatment for Atypical Endometrial Hyperplasia and Early Endometrial Cancer
Brief Title: Conservative Treatment for Atypical Endometrial Hyperplasia and Early Endometrial Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing Obstetrics and Gynecology Hospital (Other)
Responsible Party: Principal Investigator, Hongyan Ren, Researchers, Beijing Obstetrics and Gynecology Hospital
Other Study IDs: BeijingOGh，
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Atypical Endometrial Hyperplasia and Endometrial Cancer
MeSH Terms: conditions — Endometrial Hyperplasia; Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- complete remission
- non-complete remission

SUMMARY:
Exploring the efficacy and pregnancy outcomes of conservative treatment for atypical endometrial hyperplasia and endometrial cancer. Study the factors related to predicting treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

* (1) age ≤ 45 years old, strong desire to preserve reproductive function, and no factors of reproductive dysfunction evaluated before treatment; (2) The pathological type is atypical endometrial hyperplasia or endometrial cancer; (3) Imaging examination confirmed that the tumor was localized to the endometrium; (4) There are follow-up conditions available.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with atypical endometrial hyperplasia and endometrial cancer who received conservative treatment
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate | 6months